CLINICAL TRIAL: NCT06022575
Title: Evaluation of the Telehealth Integrated Care Model in Patients With Hyperlipidemia and Other Cardiometabolic Disease
Brief Title: Telehealth Integrated Care Model in Patients With Cardiometabolic Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Zeng Lin, Ph. D., Deputy Director of Research Center of Clinical Epidemiology, Peking University Third Hospital
Other Study IDs: PekingUTH Telehealth
Record Dates: First submitted 2023-07-07; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Cardiometabolic Disease; Hyperlipidemia
Keywords: Telehealth; Cardiometabolic Disease; Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Telehealth Integrated Care Group: Followed up in online Internet hospital, estimated and adjusted treatment accroding to clinical efficacy, and send individualized health education messages regularly.
  Interventions: Procedure: Telehealth integrated care
- Conventional Group: Followed up face-to-face in cardiacmetabolic clinics, estimated and adjusted treatment accroding to clinical efficacy, and conducted health education.
  Interventions: Procedure: Conventional health care

INTERVENTIONS:
Procedure: Telehealth integrated care — Followed up in online Internet hospital, estimated and adjusted treatment accroding to clinical efficacy, and send individualized health education messages regularly.
  Groups: Telehealth Integrated Care Group
Procedure: Conventional health care — Followed up face-to-face in cardiacmetabolic clinics, estimated and adjusted treatment accroding to clinical efficacy, and conducted health education.
  Groups: Conventional Group

SUMMARY:
The objective of this study is to evaluate the telehealth integrated care model for its clinical efficacy, medical resource utilization, health economics measurement, and satisfaction survey indicators in hyperlipidemia patients and other cardiometabolic diseases. The result of the study will provide evidence for the value of integrated model in the treatment of patients with cardiometabolic syndrome.

DETAILED DESCRIPTION:
Efficacy evaluation is critical for understanding the practical application effect of telehealth integrated mode in the therapy of cardiometabolic disease patients. We can comprehend the influence of the combination of online and offline models on patients' clinical curative effect, medication compliance, medical cost, and satisfaction by analyzing the curative effect and finding a scientific basis for clinical practice and policy formation. As a result, the purpose of this study is to assess the curative effect of hyperlipidemia patients with other cardiometabolic disease using a telehealth integrated model, as well as to investigate the potential benefits and risks of this model in the management of cardiometabolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years, and ≤ 85 years;
* Diagnosis as hyperlipidemia with at least one of the following disease: hypertension or type 2 diabetes mellitus;
* Agreed to be enrolled in this study.

Exclusion Criteria:

* Undergone percutaneous coronary intervention within one year in our hospital;
* Severe LV dysfunction, such as LV ejection fraction < 35%, or congestive heart failure with New York Heart Association (NYHA) functional class IV or Killip class IV;
* Structural heart disease, or severe arrhythmia;
* Severe liver or kidney diseases, endocrinology diseases, hematologic diseases, rheumatic immune system diseases, and malignancy;
* could not complete at least one-year-followup.

Ages: 16 Years to 85 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Cardiometabolic Disease
Sampling Method: Non-Probability Sample
Enrollment: 1302 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
changes of compliance rate of target treatment for hyperlipidemia | 12 month after recuitment
  difference of compliance rate of target treatment for hyperlipidemia between endpoint with baseline

SECONDARY OUTCOMES:
changes of blood pressure | 12 month after recuitment
  difference of blood pressure（both systolic and diastolic blood pressure will be measured.） between endpoint with baseline
changes of glycosylated hemoglobin | 12 month after recuitment
  difference of glycosylated hemoglobin between endpoint with baseline
changes of fasting glucose | 12 month after recuitment
  difference of fasting glucose between endpoint with baseline
changes of LDL-c | 12 month after recuitment
  difference of LDL-c between endpoint with baseline
changes of triglyceride | 12 month after recuitment
  difference of triglyceride between endpoint with baseline
abnormal liver function | 12 month after recuitment
  an increase above the 3-fold normal value for ALT or AST.
abnormal kidney function | 12 month after recuitment
  an increase in creatinine of ≥ 30%
Rehospitalization | 12 month
  Rehospitalization because of coronary heart disease, poor blood pressure control, and poor glycemic control
Cardiovascular death | 12 month
  Death because of cardiovascular diseases and sudden death
medication adherence rate | 12 month
  Difference of medication adherence between each group measured by Morisky Medication Adherence Scale-8
patients satisfaction | 12 month
  patients will be asked to rate their satisfaction score in Likert form with 1 being the most unsatisfactory and 5 being the most satisfactory on the overall experience, the medical diagnosis process, service attitude and physician's professionalism.
medical cost | 12 month
  Health Economics on medical cost, transportation cost, accommodation cost, waiting time and lost work time
in person visit counts | 12 month after recuitment
  total number of in person visits
telehealth visit counts | 12 month after recuitment
  total number of telehealth visits

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zeng, Ph.D, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided